CLINICAL TRIAL: NCT00477984
Title: The Effects of Five Dosages of Ethanol on Simulated Driving Performance and Event-Related Potentials
Brief Title: Effects of Alcohol on Simulated Driving
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Utrecht Institute for Pharmaceutical Sciences (Other)
Responsible Party: Joris Verster, Utrecht University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 06-221/O
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Last update posted 2008-04-15 (Estimated); Status verified 2008-04

CONDITIONS: Alcoholism
Keywords: Alcohol; Driving; Multitasking; ERP; social drinkers
MeSH Terms: conditions — Alcoholism | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): alcohol and placebo
  Interventions: Drug: alcohol

INTERVENTIONS:
Drug: alcohol — alcohol(0.02%, 0.05%, 0.08% and 0.10%) and placebo
  Other Names: alcohol(0.02%, 0.05%, 0.08% and 0.10%) and placebo

SUMMARY:
Previous studies have shown that alcohol significantly impairs driving performance. Acute alcohol administration also has a detrimental effect on secondary task performance during dual-tasks. The present study will investigate the effects of five different dosages of ethanol (0,0.2, 0,5, 0,8 and 1,0 % BAC) on performance in a driving simulator. Steering performance and brain activity will be recorded in both single- and dual-task conditions.

ELIGIBILITY:
Inclusion Criteria:

* He/she is aged between 21-50
* Written informed consent
* Right-handed
* Normal static binocular acuity, corrected or uncorrected
* Normal hearing
* Social Drinker (average of 7 to 21 alcoholic drinks per week)
* Possession of a drivers license
* Be considered as reliable and mentally capable of adhering to the protocol.

Exclusion Criteria:

* Current drug use (positive urine drug screen on the presence of amphetamines (including MDMA), barbiturates, cannabinoids, benzodiazepines, cocaine, and opiates)
* Positive urine pregnancy drug screen in women
* Use of psychoactive medication
* Positive alcohol breath test
* Prior enrolment in the same study
* Physical or mental illness
* Excessive alcohol use (>21 alcoholic drinks per week)
* Excessive smoking (more than 10 cigarettes per day)
* Intake of caffeine-containing beverages over 5 glasses per day

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2007-05; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Primary parameter of the steering simulator is the standard deviation of the car from the center of the road (steering error). | 5 testdays

SECONDARY OUTCOMES:
Reaction speed after hearing the deviant target tone. Brain activity: ERPs of interest are the mismatch negativity (MMN), P3a, P3b, and reorienting negativity (RON) | 5 testdays

CONTACTS AND LOCATIONS:
Overall Officials: Joris C Verster, PhD, Principal Investigator — Utrecht Institute for Pharmaceutical Sciences; Edmund R Volkerts, PhD, Study Director — Utrecht Institute for Pharmaceutical Sciences
Locations (1):
- Utrecht Institute for Pharmaceutical Sciences, Utrecht, Utrecht, Netherlands